CLINICAL TRIAL: NCT06001788
Title: Phase 1 Study to Determine the Safety and Tolerability of Ziftomenib Combinations for the Treatment of KMT2A-rearranged or NPM1-mutant Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Safety and Tolerability of Ziftomenib Combinations in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KO-MEN-008
Expanded Access: NCT05738538 (Available)
Record Dates: First submitted 2023-08-07; First posted 2023-08-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: AML; AML With Mutated NPM1; Hematologic Malignancy; KMT2Ar; NPM1 Mutation; MLL Rearrangement; Leukemia; Acute Myeloid Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute; Acute Leukemia; Neoplasms by Histologic Type
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Leukemia, Myeloid, Acute; Leukemia, Myeloid; Neoplasms by Histologic Type | interventions — fludarabine; Idarubicin; Cytarabine; gilteritinib; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a (Experimental): Oral ziftomenib; sequential cohorts of escalating dose levels of ziftomenib to identify the safety and tolerability of the combination regimens. Participants will be enrolled in 1 of 5 dose escalation cohorts:
  A-1: Participants with a NPM1 mutation: ziftomenib plus FLAG-IDA
  A-2: Participants with a NPM1 mutation: ziftomenib plus low-dose cytarabine (LDAC)
  A-3: Participants with a NPM1 mutation: ziftomenib plus gilteritinib
  B-1: Participants with a KMT2A rearrangement: ziftomenib plus FLAG-IDA
  B-2: Participants with a KMT2A rearrangement: ziftomenib plus low-dose cytarabine (LDAC)
  Interventions: Drug: Ziftomenib; Drug: Fludarabine; Drug: Idarubicin; Drug: Cytarabine; Drug: Gilteritinib; Biological: Granulocyte colony-stimulating factor
- Phase 1b (Experimental): Oral ziftomenib; Following the determination of the maximum tolerated dose in Phase 1a, participants will be enrolled in 1 of 5 dose validation/expansion cohorts:
  A-1: Participants with a NPM1 mutation: ziftomenib plus FLAG-IDA
  A-2: Participants with a NPM1 mutation: ziftomenib plus low-dose cytarabine (LDAC)
  A-3: Participants with a NPM1 mutation: ziftomenib plus gilteritinib
  B-1: Participants with a KMT2A rearrangement: ziftomenib plus FLAG-IDA
  B-2: Participants with a KMT2A rearrangement: ziftomenib plus low-dose cytarabine (LDAC)
  Interventions: Drug: Ziftomenib; Drug: Fludarabine; Drug: Idarubicin; Drug: Cytarabine; Drug: Gilteritinib; Biological: Granulocyte colony-stimulating factor

INTERVENTIONS:
Drug: Ziftomenib — Oral administration
  Other Names: KO-539
Drug: Fludarabine — Intravenous infusion
Drug: Idarubicin — Intravenous infusion
Drug: Cytarabine — Intravenous Infusion
Drug: Gilteritinib — Oral administration
  Other Names: Xospata
Biological: Granulocyte colony-stimulating factor — Subcutaneous injection

SUMMARY:
The safety, tolerability, and antileukemic response of ziftomenib in combination with standard of care treatments for patients with relapsed/refractory acute myeloid leukemia will be examined with the following agents: FLAG-IDA, low-dose cytarabine, and gilteritinib.

ELIGIBILITY:
Key Inclusion Criteria:

* Has been diagnosed with relapsed/refractory AML.
* Has a documented NPM1 mutation or KMT2A rearrangement.
* Has a documented FLT3 mutation (cA-3 only).
* Has an Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2.
* Has adequate hepatic and renal function as defined per protocol.
* Has an ejection fraction above a protocol defined limit.
* Participant, or legally authorized representative, must be able to understand and provide written informed consent prior to the first screening procedure.
* Has agreed to use contraception as defined per protocol.

Key Exclusion Criteria:

* Has a diagnosis of acute promyelocytic leukemia or blast chronic myeloid leukemia.
* Has clinically active central nervous system leukemia.
* Has an active and uncontrolled infection.
* Has a mean corrected QT interval (QTcF) > 480ms.
* Has uncontrolled intercurrent illness, including, but not limited to protocol defined cardiac disease.
* Has received radiation, chemotherapy, immunotherapy, or any other anticancer therapy including investigational therapy <14 days or within 5 drug half-lives prior to the first dose of study intervention.
* Has had major surgery within 4 weeks prior to the first dose of study intervention.
* Has received a hematopoietic stem cell transplant (HSCT) and has not previously had adequate recovery per protocol defined criteria.
* Has active graft-versus-host disease (GvHD) and or on immunosuppressive drugs for the treatment of GvHD
* Participant is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities (DLTs) per dose level | During the first 28 days of ziftomenib in combination with SOC treatment (1 cycle)
  Assessed by the NCI-CTCAE v5.0
Descriptive statistics of adverse events | First dose of ziftomenib up to and including 28 days after last dose of ziftomenib, or if the patient is lost to follow-up, whichever comes first
  Assessed by the NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Complete remission (CR) rate for cohorts A-1, A-2, B-1, and B-2 | Up to 12 months following discontinuation of treatment
  Assessed by ELN 2022 criteria
Complete remission (CR) / Complete remission with partial hematologic recovery (CRh) rate for cohort A-3 | Up to 12 months following discontinuation of treatment
  Assessed by ELN 2022 criteria
Composite complete remission (CRc) rate | Up to 12 months following discontinuation of treatment
  Assessed by ELN 2022 criteria
Morphologic leukemia-free state (MLFS) rate | Up to 12 months following discontinuation of treatment
  Assessed by ELN 2022 criteria
OS | Up to 12 months following discontinuation of treatment
  To assess overall survival
6-month OS | Up to 6 months following discontinuation of treatment
  To assess proportion of patients alive at 6 months
Median EFS | Up to 12 months following discontinuation of treatment
  To assess median event free survival
6-month EFS | Up to 6 months following discontinuation of treatment
  To assess 6-month event free survival
DOR | Up to 12 months following discontinuation of treatment
  To assess duration of remission
MRD assessment | Up to 12 months following discontinuation of treatment
  To assess minimum residual disease in bone marrow as assessed by multiparameter flow cytometry (MFC) and molecular analysis
HSCT | Up to 12 months following discontinuation of treatment
  To assess proportion of patients that undergo a hematopoietic stem-cell transplant
Transfusion independence | Up to 12 months following discontinuation of treatment
  To assess rate of transfusion independence
Ziftomenib Cmax | Cycle 1 (Each cycle is 28 days)
  To assess the maximum plasma combination of ziftomenib and its metabolites
Ziftomenib Tmax | Cycle 1 (Each cycle is 28 days)
  To assess the time to observed maximum plasma concentration of ziftomenib and its metabolites
Ziftomenib AUC(0-last) | Cycle 1 (Each cycle is 28 days)
  To assess the area under the plasma concentration-time-curve from time 0 to time of last measurable concentration of ziftomenib and its metabolites
Ziftomenib AUC(tau) | Cycle 1 (Each cycle is 28 days)
  To assess the area under the plasma concentration-time-curve over a dosing interval for ziftomenib and its metabolites
Gilteritinib Cmax | Cycle 1 (Each cycle is 28 days)
  To assess the maximum plasma combination of gilteritinib
Gilteritinib Tmax | Cycle 1 (Each cycle is 28 days)
  To assess the time to observed maximum plasma concentration of gilteritinib
Gilteritinib AUC(0-last) | Cycle 1 (Each cycle is 28 days)
  To assess the area under the plasma concentration-time-curve from time 0 to time of last measurable concentration of gilteritinib
Gilteritinib AUC(tau) | Cycle 1 (Each cycle is 28 days)
  To assess the area under the plasma concentration-time-curve over a dosing interval for gilteritinib

CONTACTS AND LOCATIONS:
Locations (44):
- United States (37):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Health - Bowyer Oncology Center, Los Angeles, California
  - UC Irvine Health Chao Family Comprehensive Cancer Center, Orange, California
  - University of California San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Emory Healthcare - The Emory Clinic, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Simmons Cancer Institute, Springfield, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - The University of Kansas Cancer Center, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Cancer Institute, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Northwell Health, LLC PRIME, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College-NY Presbyterian Hospital, New York, New York
  - Wilmot Cancer Institute, University of Rochester, Rochester, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Atrium Health Levine Cancer Center, Charlotte, North Carolina
  - UH Seidman Cancer Center, Cleveland, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Lehigh Valley Topper Cancer Institute, Allentown, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Vermont, Burlington, Vermont
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
  - Froedtert & Medical College Clinics, Milwaukee, Wisconsin
- Italy (3):
  - IRCCS Azienda Ospedaliero-Universitaria do Bologna - Policlinico di Sant'Orsola, Bologna
  - Ospedale Santa Maria delle Croci, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari y Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided